CLINICAL TRIAL: NCT06401330
Title: Risk Adapted Treatment of Unilateral Favorable Histology Wilms Tumors (FHWT)
Brief Title: A Study Using Risk Factors to Determine Treatment for Children With Favorable Histology Wilms Tumors (FHWT)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AREN2231; NCI-2024-03424 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AREN2231 (Other: Children's Oncology Group); AREN2231 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Stage I Mixed Cell Type Kidney Wilms Tumor; Stage II Mixed Cell Type Kidney Wilms Tumor; Stage III Mixed Cell Type Kidney Wilms Tumor; Stage IV Mixed Cell Type Kidney Wilms Tumor
MeSH Terms: interventions — Carboplatin; Cyclophosphamide; Dactinomycin; Doxorubicin; Etoposide; Irinotecan; Magnetic Resonance Spectroscopy; Nephrectomy; Watchful Waiting; Observation; High-Energy Shock Waves; Vincristine; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (48):
- Stage I, Arm I (EE-4A) (Experimental): Patients receive regimen EE-4A: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycles 1-7 and vincristine IV on days 1, 8, & 15 of cycles 1-3 and day 1 of cycles 4-7. Treatment repeats every 21 days for 7 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Biological: Dactinomycin; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage I, Arm II (observation) (Experimental): Patients undergo observation without chemotherapy on study with ultrasounds and x-rays.
  Interventions: Other: Patient Observation; Procedure: Ultrasound Imaging; Procedure: X-Ray Imaging
- Stage I, Arm III (DD-4A) (Experimental): Patients receive regimen DD-4A: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycles 1, 3, 5, 7, & 9, vincristine IV on days 1, 8, & 15 of cycles 1-3 and day 1 of cycles 4-9, doxorubicin IV over 3-15 minutes on day 1 of cycles 2, 4, 6, & 8. Treatment repeats every 21 days for 9 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Biological: Dactinomycin; Drug: Doxorubicin; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage I, Arm IV (UH-3) (Experimental): Patients receive regimen UH-3: Vincristine IV on days 1, 8, & 15 of cycles 1, 5, 7, 10, & 13, and days 1 & 8 of cycles 3, 4, 8, & 11, doxorubicin IV 3-15 minutes on day 1 of cycles 1, 5, 7, 10, & 13, cyclophosphamide IV over 30-60 minutes on day 1 of cycles 1, 5, 7, 10, & 13, and days 1-4 of cycles 2, 6, 9, 12, & 14, carboplatin IV over 15-60 minutes on day 1 of cycles 2, 6, 9, 12, and 14, etoposide IV over 60-120 minutes on days 1-4 of cycles 2, 6, 9, 12, & 14, and irinotecan IV over 90 minutes on days 1-5 of cycles 3, 4, 8, & 11. Treatment repeats every 21 days for 14 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Drug: Carboplatin; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage II, Arm I (EE-4A) (Experimental): Patients receive one cycle of regimen EE-4A as in STAGE I FHWT Arm I. Patients receive cycles 2-7 of regimen EE-4A as in STAGE I FHWT Arm I. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Biological: Dactinomycin; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage II, Arm II (EE-4A, VIVA) (Experimental): Patients receive one cycle of regimen EE-4A as in STAGE I FHWT Arm I. Patients receive cycles 2-9 of regimen VIVA: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycles 3, 5, 7, & 9, vincristine IV on days 1, 8, & 15 of cycles 2-3 and day 1 of cycles 4-9, irinotecan IV over 90 minutes daily on days 1-5 of cycles 2, 4, 6, & 8. Treatment repeats every 21 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Biological: Dactinomycin; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage II, Arm III (EE-4A, DD-4A) (Experimental): Patients receive one cycle of regimen EE-4A as in STAGE I FHWT Arm I. Patients receive cycles 2-9 of regimen DD-4A: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycles 3, 5, 7, and 9, vincristine IV on days 1, 8, and 15 of cycles 2-3 and day 1 of cycles 4-9, and doxorubicin IV over 3-15 minutes on day 1 of cycles 2, 4, 6, & 8. Treatment repeats every 21 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Biological: Dactinomycin; Drug: Doxorubicin; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage III, Arm I (DD-4A, EE-4A) (Experimental): Patients able to undergo an upfront nephrectomy receive cycle 1 treatment of regimen DD-4A: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycles 1, 3, 5, 7, & 9, vincristine IV on days 1, 8, & 15 of cycles 1-3 and day 1 of cycles 4-9, doxorubicin IV over 3-15 minutes on day 1 of cycles 2, 4, 6, & 8. Patients with standard biology receive cycles 2-7 of regimen EE-4A as in STAGE I FHWT Arm I. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Biological: Dactinomycin; Drug: Doxorubicin; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage III, Arm I-Upfront/Delayed (DD-4A, EE-4A) (Experimental): Patients receive cycles 1-2 of regimen DD-4A: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycle 1, vincristine IV on days 1, 8, and 15 of cycles 1-2, and doxorubicin IV over 3-15 minutes on day 1 of cycle 2. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients receive cycles 3-7 of regimen EE-4A as in STAGE I FHWT Arm I above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Biological: Dactinomycin; Drug: Doxorubicin; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage III, Arm II (DD-4A) (Experimental): Patients able to undergo an upfront nephrectomy receive cycle 1 treatment of regimen DD-4A: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycles 1, 3, 5, 7, & 9, vincristine IV on days 1, 8, & 15 of cycles 1-3 and day 1 of cycles 4-9, doxorubicin IV over 3-15 minutes on day 1 of cycles 2, 4, 6, & 8. Patients with adverse biology receive cycle 2 treatment of regimen DD-4A as in STAGE II FHWT Arm III above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Biological: Dactinomycin; Drug: Doxorubicin; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage III, Arm II-Upfront/Delayed (DD-4A, UH-3) (Experimental): Patients receive cycles 1-2 of regimen DD-4A: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycle 1, vincristine IV on days 1, 8, and 15 of cycles 1-2, and doxorubicin IV over 3-15 minutes on day 1 of cycle 2. Patients receive regimen UH-3 as in STAGE I FHWT Arm IV above: Vincristine IV on days 1, 8, & 15 of cycles 1, 5, 7, 10, & 13, and days 1 & 8 of cycles 3, 4, 8, & 11, doxorubicin IV 3-15 minutes on day 1 of cycles 1, 5, 7, 10, & 13, cyclophosphamide IV over 30-60 minutes on day 1 of cycles 1, 5, 7, 10, & 13, and days 1-4 of cycles 2, 6, 9, 12, & 14, carboplatin IV over 15-60 minutes on day 1 of cycles 2, 6, 9, 12, and 14, etoposide IV over 60-120 minutes on days 1-4 of cycles 2, 6, 9, 12, & 14, and irinotecan IV over 90 minutes on days 1-5 of cycles 3, 4, 8, & 11. Treatment repeats every 21 days for 14 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Drug: Carboplatin; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage III, Arm IIA (MVI) (Experimental): Patients receive regimen MVI: Vincristine IV on days 1, 8, & 15 of cycle 3, days 8 & 15 of cycle 4, and day 1 of cycles 5 & 7-13, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycles 3, 7, 9, 11, & 13, doxorubicin IV over 3-15 minutes on day 1 of cycles 3, 7, 9, 11, & 13, cyclophosphamide IV over 15-30 minutes daily on days 1-5 of cycles 4 and 6, irinotecan IV over 90 minutes daily on days 1-5 of cycles 5, 8, 10 & 12, and etoposide IV over 60-120 minutes daily on days 1-5 of cycles 4 and 6. Treatment repeats every 21 days for 11 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage III, Arm IIB (M) (Experimental): Patients receive regimen M: Cyclophosphamide IV over 15-30 minutes daily on days 1-5 of cycles 3, 4, 7, & 9, etoposide IV over 60-120 minutes daily on days 1-5 of cycles 3, 4, 7, & 9, vincristine IV on days 8 & 15 of cycles 3 & 4 and day 1 of cycles 5, 6, 8, 10, & 11, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycles 5, 6, 8, 10, & 11, and doxorubicin IV over 3-15 minutes of cycles 5, 6, 8, 10, & 11. Treatment repeats every 21 days for 9 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage III, Arm III-Upfront/Delayed (DD-4A, MVI) (Experimental): Patients receive cycles 1-2 of regimen DD-4A: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycle 1, vincristine IV on days 1, 8, and 15 of cycles 1-2, and doxorubicin IV over 3-15 minutes on day 1 of cycle 2. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients receive regimen MVI as in STAGE III FHWT Arm IIA above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage III, Arm IV-Upfront/Delayed (DD-4A, M) (Experimental): Patients receive cycles 1-2 of regimen DD-4A: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycle 1, vincristine IV on days 1, 8, and 15 of cycles 1-2, and doxorubicin IV over 3-15 minutes on day 1 of cycle 2. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients receive regimen M as in STAGE III FHWT Arm IIB above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage III, Arm IX-Upfront/Delayed (MVI) (Experimental): Patients receive cycles 5-13 (or 4-13 if nephrectomy occurred after cycle 3) of regimen MVI as in STAGE III FHWT Arm IIA above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage III, Arm V-Upfront/Delayed (DD-4A) (Experimental): Patients receive cycles 1-2 of regimen DD-4A: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycle 1, vincristine IV on days 1, 8, and 15 of cycles 1-2, and doxorubicin IV over 3-15 minutes on day 1 of cycle 2. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients receive cycles 3-4 of regimen DD-4A as in STAGE II FHWT Arm III above. They then undergo delayed nephrectomy after cycle 3 or 4. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Biological: Dactinomycin; Drug: Doxorubicin; Procedure: Magnetic Resonance Imaging; Procedure: Nephrectomy; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage III, Arm VA-Upfront/Delayed (DD-4A) (Experimental): Patients receive cycles 5-9 (or 4-9 if nephrectomy occurred after cycle 3) of regimen DD-4A as in STAGE II FHWT Arm III above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Biological: Dactinomycin; Drug: Doxorubicin; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage III, Arm VB-Upfront/Delayed (M) (Experimental): Patients receive cycles 5-9 (or 4-9 if nephrectomy occurred after cycle 3) of regimen M as in STAGE III FHWT Arm IIB above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Procedure: X-Ray Imaging
- Stage III, Arm VI-Upfront/Delayed (DD-4A, MVI) (Experimental): Patients receive cycles 1-2 of regimen DD-4A: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycle 1, vincristine IV on days 1, 8, and 15 of cycles 1-2, and doxorubicin IV over 3-15 minutes on day 1 of cycle 2. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients receive cycles 3-4 of regimen MVI as in STAGE III FHWT Arm IIA above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage III, Arm VII-Upfront/Delayed (DD-4A, M) (Experimental): Patients receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive cycles 3-4 of regimen M as in STAGE III FHWT Arm IIB above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage III, Arm VIII-Upfront/Delayed (UH-3) (Experimental): Patients receive regimen UH-3 as in STAGE I FHWT Arm IV above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Drug: Carboplatin; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage III, Arm X-Upfront/Delayed (M) (Experimental): Patients receive cycles 5-11 (or 4-11 if nephrectomy occurred after cycle 3) of regimen M as in STAGE III FHWT Arm IIB above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Arm I-Upfront-Delayed (DD-4A, EE-4A) (Experimental): Patients receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive cycles 3-7 of regimen EE-4A as in STAGE I FHWT Arm I above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Biological: Dactinomycin; Drug: Doxorubicin; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Arm II-Upfront-Delayed (DD-4A, UH-3) (Experimental): Patients receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive regimen UH-3 as in STAGE I FHWT Arm IV above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Drug: Carboplatin; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Arm III-Upfront-Delayed (DD-4A, MVI) (Experimental): Patients in Stage IV Arm III Upfront-Delayed receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive regimen MVI as in STAGE III FHWT Arm IIA above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Arm IV-Upfront-Delayed (DD-4A, M) (Experimental): Patients in Stage IV Arm IV Upfront-Delayed receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive regimen M as in STAGE III FHWT Arm IIB above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Arm IX-Upfront-Delayed (MVI) (Experimental): Patients in Stage IV Arm IX Upfront-Delayed receive cycles 5-13 (or 4-13 if nephrectomy occurred after cycle 3) of regimen MVI as in STAGE III FHWT Arm IIA above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Arm V-Upfront-Delayed (DD-4A) (Experimental): Patients receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive cycles 3-4 of regimen DD-4A as in STAGE II FHWT Arm II above. They then undergo delayed nephrectomy after cycle 3 or 4. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Biological: Dactinomycin; Drug: Doxorubicin; Procedure: Magnetic Resonance Imaging; Procedure: Nephrectomy; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Arm VA-Upfront-Delayed (DD-4A) (Experimental): Patients receive cycles 5-9 (or 4-9 if nephrectomy occurred after cycle 3) of regimen DD-4A as in STAGE II FHWT Arm II above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Biological: Dactinomycin; Drug: Doxorubicin; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Arm VB-Upfront-Delayed (M) (Experimental): Patients receive regimen M as in STAGE III FHWT Arm IIB above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Arm VI-Upfront-Delayed (DD-4A, MVI) (Experimental): Patients receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive cycles 3-4 of regimen MVI as in STAGE III FHWT Arm IIA above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Arm VII-Upfront-Delayed (DD-4A, M) (Experimental): Patients in Stage IV Arm VII Upfront-Delayed receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive cycles 3-4 of regimen M as in STAGE III FHWT Arm IIB above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Arm VIII-Upfront-Delayed (UH-3) (Experimental): Patients in Stage IV Arm VIII Upfront-Delayed receive regimen UH-3 as in STAGE I FHWT Arm IV above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Drug: Carboplatin; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Arm X-Upfront-Delayed (M) (Experimental): Patients receive cycles 5-11 (or 4-11 if nephrectomy occurred after cycle 3) of regimen M as in STAGE III FHWT Arm IIB above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Extrapulmonary Arm I (DD-4A, MVI) (Experimental): Patients in Stage IV Extrapulmonary Arm I receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive regimen MVI as in STAGE III FHWT Arm IIA above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial. Patients with metastatic sites outside the chest/abdomen/pelvis documented during therapy may undergo bone scan and/or PET.
  Interventions: Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Extrapulmonary Arm II (DD-4A, M) (Experimental): Patients in Stage IV Extrapulmonary Arm II receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive regimen M as in STAGE III FHWT Arm IIB above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial. Patients with metastatic sites outside the chest/abdomen/pelvis documented during therapy may undergo bone scan and/or PET.
  Interventions: Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Extrapulmonary Arm III (DD-4A, MVI) (Experimental): Patients in Stage IV Extrapulmonary Arm III receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive regimen MVI as in STAGE III FHWT Arm IIA above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial. Patients with metastatic sites outside the chest/abdomen/pelvis documented during therapy may undergo bone scan and/or PET.
  Interventions: Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Extrapulmonary Arm IV (DD-4A, M) (Experimental): Patients in Stage IV Extrapulmonary Arm IV receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive regimen M as in STAGE III FHWT Arm IIB above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial. Patients with metastatic sites outside the chest/abdomen/pelvis documented during therapy may undergo bone scan and/or PET.
  Interventions: Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Extrapulmonary Arm IX (MVI) (Experimental): Patients in Stage IV Extrapulmonary Arm IX receive cycles 5-13 (or 4-13 if nephrectomy occurred after cycle 3) of regimen MVI as in STAGE III FHWT Arm IIA above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial. Patients with metastatic sites outside the chest/abdomen/pelvis documented during therapy may undergo bone scan and/or PET.
  Interventions: Procedure: Bone Scan; Procedure: Computed Tomography; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Extrapulmonary Arm V (DD-4A, UH-3) (Experimental): Patients receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive regimen UH-3 as in STAGE I FHWT Arm IV above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial. Patients with metastatic sites outside the chest/abdomen/pelvis documented during therapy may undergo bone scan and/or PET.
  Interventions: Procedure: Bone Scan; Drug: Carboplatin; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Extrapulmonary Arm VI (DD-4A, MVI) (Experimental): Patients in Stage IV Extrapulmonary Arm VI receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive cycles 3-4 of regimen MVI as in STAGE III FHWT Arm IIA above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial. Patients with metastatic sites outside the chest/abdomen/pelvis documented during therapy may undergo bone scan and/or PET.
  Interventions: Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Extrapulmonary Arm VII (DD-4A, M) (Experimental): Patients in Stage IV Extrapulmonary Arm VII receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive cycles 3-4 of regimen M as in STAGE III FHWT Arm IIB above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial. Patients with metastatic sites outside the chest/abdomen/pelvis documented during therapy may undergo bone scan and/or PET.
  Interventions: Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Extrapulmonary Arm VIII (UH-3) (Experimental): Patients in Stage IV Extrapulmonary Arm VIII receive regimen UH-3 as in STAGE I FHWT Arm IV above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial. Patients with metastatic sites outside the chest/abdomen/pelvis documented during therapy may undergo bone scan and/or PET.
  Interventions: Procedure: Bone Scan; Drug: Carboplatin; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Extrapulmonary Arm X (M) (Experimental): Patients in Stage IV Extrapulmonary Arm X receive cycles 5-11 (or 4-11 if nephrectomy occurred after cycle 3) of regimen M as in STAGE III FHWT Arm IIB above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial. Patients with metastatic sites outside the chest/abdomen/pelvis documented during therapy may undergo bone scan and/or PET.
  Interventions: Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Lung Metastases Arm I (DD-4A) (Experimental): Patients receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive cycles 3-9 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) Arms V and VA above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Biological: Dactinomycin; Drug: Doxorubicin; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Lung Metastases Arm II (DD-4A, MVI) (Experimental): Patients receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive regimen MVI as in STAGE III FHWT Arm IIA above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Drug: Irinotecan; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging
- Stage IV Lung Metastases Arm III (DD-4A, MVI) (Experimental): Patients receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients receive regimen M as in STAGE III FHWT Arm IIB above. Patients also undergo CT, CT or MRI, ultrasound, and X-ray imaging throughout the trial.
  Interventions: Procedure: Computed Tomography; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Drug: Vincristine; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Bone Scan — Undergo bone scan for patients with metastatic sites outside the chest/abdomen/pelvis documented during therapy
  Other Names: Bone Scintigraphy
  Arms: Stage III, Arm IIA (MVI); Stage IV Arm VI-Upfront-Delayed (DD-4A, MVI); Stage IV Arm X-Upfront-Delayed (M); Stage IV Extrapulmonary Arm I (DD-4A, MVI); Stage IV Extrapulmonary Arm II (DD-4A, M); Stage IV Extrapulmonary Arm III (DD-4A, MVI); Stage IV Extrapulmonary Arm IV (DD-4A, M); Stage IV Extrapulmonary Arm IX (MVI); Stage IV Extrapulmonary Arm V (DD-4A, UH-3); Stage IV Extrapulmonary Arm VI (DD-4A, MVI); Stage IV Extrapulmonary Arm VII (DD-4A, M); Stage IV Extrapulmonary Arm VIII (UH-3); Stage IV Extrapulmonary Arm X (M)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Stage I, Arm IV (UH-3); Stage III, Arm II-Upfront/Delayed (DD-4A, UH-3); Stage III, Arm VIII-Upfront/Delayed (UH-3); Stage IV Arm II-Upfront-Delayed (DD-4A, UH-3); Stage IV Arm VIII-Upfront-Delayed (UH-3); Stage IV Extrapulmonary Arm V (DD-4A, UH-3); Stage IV Extrapulmonary Arm VIII (UH-3)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
  Arms: Stage I, Arm I (EE-4A); Stage I, Arm III (DD-4A); Stage I, Arm IV (UH-3); Stage II, Arm I (EE-4A); Stage II, Arm II (EE-4A, VIVA); Stage II, Arm III (EE-4A, DD-4A); Stage III, Arm I (DD-4A, EE-4A); Stage III, Arm I-Upfront/Delayed (DD-4A, EE-4A); Stage III, Arm II (DD-4A); Stage III, Arm II-Upfront/Delayed (DD-4A, UH-3); Stage III, Arm IIA (MVI); Stage III, Arm IIB (M); Stage III, Arm III-Upfront/Delayed (DD-4A, MVI); Stage III, Arm IV-Upfront/Delayed (DD-4A, M); Stage III, Arm IX-Upfront/Delayed (MVI); Stage III, Arm V-Upfront/Delayed (DD-4A); Stage III, Arm VA-Upfront/Delayed (DD-4A); Stage III, Arm VB-Upfront/Delayed (M); Stage III, Arm VI-Upfront/Delayed (DD-4A, MVI); Stage III, Arm VII-Upfront/Delayed (DD-4A, M); Stage III, Arm VIII-Upfront/Delayed (UH-3); Stage III, Arm X-Upfront/Delayed (M); Stage IV Arm I-Upfront-Delayed (DD-4A, EE-4A); Stage IV Arm II-Upfront-Delayed (DD-4A, UH-3); Stage IV Arm III-Upfront-Delayed (DD-4A, MVI); Stage IV Arm IV-Upfront-Delayed (DD-4A, M); Stage IV Arm IX-Upfront-Delayed (MVI); Stage IV Arm V-Upfront-Delayed (DD-4A); Stage IV Arm VA-Upfront-Delayed (DD-4A); Stage IV Arm VB-Upfront-Delayed (M); Stage IV Arm VI-Upfront-Delayed (DD-4A, MVI); Stage IV Arm VII-Upfront-Delayed (DD-4A, M); Stage IV Arm VIII-Upfront-Delayed (UH-3); Stage IV Arm X-Upfront-Delayed (M); Stage IV Extrapulmonary Arm I (DD-4A, MVI); Stage IV Extrapulmonary Arm II (DD-4A, M); Stage IV Extrapulmonary Arm III (DD-4A, MVI); Stage IV Extrapulmonary Arm IV (DD-4A, M); Stage IV Extrapulmonary Arm IX (MVI); Stage IV Extrapulmonary Arm V (DD-4A, UH-3); Stage IV Extrapulmonary Arm VI (DD-4A, MVI); Stage IV Extrapulmonary Arm VII (DD-4A, M); Stage IV Extrapulmonary Arm VIII (UH-3); Stage IV Extrapulmonary Arm X (M); Stage IV Lung Metastases Arm I (DD-4A); Stage IV Lung Metastases Arm II (DD-4A, MVI); Stage IV Lung Metastases Arm III (DD-4A, MVI)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
  Arms: Stage I, Arm IV (UH-3); Stage III, Arm II-Upfront/Delayed (DD-4A, UH-3); Stage III, Arm IIA (MVI); Stage III, Arm IIB (M); Stage III, Arm III-Upfront/Delayed (DD-4A, MVI); Stage III, Arm IV-Upfront/Delayed (DD-4A, M); Stage III, Arm IX-Upfront/Delayed (MVI); Stage III, Arm VB-Upfront/Delayed (M); Stage III, Arm VI-Upfront/Delayed (DD-4A, MVI); Stage III, Arm VII-Upfront/Delayed (DD-4A, M); Stage III, Arm VIII-Upfront/Delayed (UH-3); Stage III, Arm X-Upfront/Delayed (M); Stage IV Arm II-Upfront-Delayed (DD-4A, UH-3); Stage IV Arm III-Upfront-Delayed (DD-4A, MVI); Stage IV Arm IV-Upfront-Delayed (DD-4A, M); Stage IV Arm IX-Upfront-Delayed (MVI); Stage IV Arm VB-Upfront-Delayed (M); Stage IV Arm VI-Upfront-Delayed (DD-4A, MVI); Stage IV Arm VII-Upfront-Delayed (DD-4A, M); Stage IV Arm VIII-Upfront-Delayed (UH-3); Stage IV Arm X-Upfront-Delayed (M); Stage IV Extrapulmonary Arm I (DD-4A, MVI); Stage IV Extrapulmonary Arm II (DD-4A, M); Stage IV Extrapulmonary Arm III (DD-4A, MVI); Stage IV Extrapulmonary Arm IV (DD-4A, M); Stage IV Extrapulmonary Arm V (DD-4A, UH-3); Stage IV Extrapulmonary Arm VI (DD-4A, MVI); Stage IV Extrapulmonary Arm VII (DD-4A, M); Stage IV Extrapulmonary Arm VIII (UH-3); Stage IV Extrapulmonary Arm X (M); Stage IV Lung Metastases Arm II (DD-4A, MVI); Stage IV Lung Metastases Arm III (DD-4A, MVI)
Biological: Dactinomycin — Given IV
  Other Names: Actinomycin A IV; Actinomycin C1; Actinomycin D; Actinomycin I1; Actinomycin IV; Actinomycin X 1; Actinomycin-[thr-val-pro-sar-meval]; Cosmegen; DACT; Dactinomycine; Lyovac Cosmegen; Meractinomycin
  Arms: Stage I, Arm I (EE-4A); Stage I, Arm III (DD-4A); Stage II, Arm I (EE-4A); Stage II, Arm II (EE-4A, VIVA); Stage II, Arm III (EE-4A, DD-4A); Stage III, Arm I (DD-4A, EE-4A); Stage III, Arm I-Upfront/Delayed (DD-4A, EE-4A); Stage III, Arm II (DD-4A); Stage III, Arm II-Upfront/Delayed (DD-4A, UH-3); Stage III, Arm IIA (MVI); Stage III, Arm IIB (M); Stage III, Arm III-Upfront/Delayed (DD-4A, MVI); Stage III, Arm IV-Upfront/Delayed (DD-4A, M); Stage III, Arm IX-Upfront/Delayed (MVI); Stage III, Arm V-Upfront/Delayed (DD-4A); Stage III, Arm VA-Upfront/Delayed (DD-4A); Stage III, Arm VB-Upfront/Delayed (M); Stage III, Arm VI-Upfront/Delayed (DD-4A, MVI); Stage III, Arm VII-Upfront/Delayed (DD-4A, M); Stage III, Arm X-Upfront/Delayed (M); Stage IV Arm I-Upfront-Delayed (DD-4A, EE-4A); Stage IV Arm II-Upfront-Delayed (DD-4A, UH-3); Stage IV Arm III-Upfront-Delayed (DD-4A, MVI); Stage IV Arm IV-Upfront-Delayed (DD-4A, M); Stage IV Arm IX-Upfront-Delayed (MVI); Stage IV Arm V-Upfront-Delayed (DD-4A); Stage IV Arm VA-Upfront-Delayed (DD-4A); Stage IV Arm VB-Upfront-Delayed (M); Stage IV Arm VI-Upfront-Delayed (DD-4A, MVI); Stage IV Arm VII-Upfront-Delayed (DD-4A, M); Stage IV Arm X-Upfront-Delayed (M); Stage IV Extrapulmonary Arm I (DD-4A, MVI); Stage IV Extrapulmonary Arm II (DD-4A, M); Stage IV Extrapulmonary Arm IV (DD-4A, M); Stage IV Extrapulmonary Arm IX (MVI); Stage IV Extrapulmonary Arm V (DD-4A, UH-3); Stage IV Extrapulmonary Arm VI (DD-4A, MVI); Stage IV Extrapulmonary Arm VII (DD-4A, M); Stage IV Lung Metastases Arm I (DD-4A); Stage IV Lung Metastases Arm II (DD-4A, MVI); Stage IV Lung Metastases Arm III (DD-4A, MVI)
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
  Arms: Stage I, Arm III (DD-4A); Stage I, Arm IV (UH-3); Stage II, Arm III (EE-4A, DD-4A); Stage III, Arm I (DD-4A, EE-4A); Stage III, Arm I-Upfront/Delayed (DD-4A, EE-4A); Stage III, Arm II (DD-4A); Stage III, Arm II-Upfront/Delayed (DD-4A, UH-3); Stage III, Arm IIA (MVI); Stage III, Arm IIB (M); Stage III, Arm III-Upfront/Delayed (DD-4A, MVI); Stage III, Arm IV-Upfront/Delayed (DD-4A, M); Stage III, Arm IX-Upfront/Delayed (MVI); Stage III, Arm V-Upfront/Delayed (DD-4A); Stage III, Arm VA-Upfront/Delayed (DD-4A); Stage III, Arm VB-Upfront/Delayed (M); Stage III, Arm VI-Upfront/Delayed (DD-4A, MVI); Stage III, Arm VII-Upfront/Delayed (DD-4A, M); Stage III, Arm VIII-Upfront/Delayed (UH-3); Stage III, Arm X-Upfront/Delayed (M); Stage IV Arm I-Upfront-Delayed (DD-4A, EE-4A); Stage IV Arm II-Upfront-Delayed (DD-4A, UH-3); Stage IV Arm III-Upfront-Delayed (DD-4A, MVI); Stage IV Arm IV-Upfront-Delayed (DD-4A, M); Stage IV Arm IX-Upfront-Delayed (MVI); Stage IV Arm V-Upfront-Delayed (DD-4A); Stage IV Arm VA-Upfront-Delayed (DD-4A); Stage IV Arm VB-Upfront-Delayed (M); Stage IV Arm VI-Upfront-Delayed (DD-4A, MVI); Stage IV Arm VII-Upfront-Delayed (DD-4A, M); Stage IV Arm VIII-Upfront-Delayed (UH-3); Stage IV Arm X-Upfront-Delayed (M); Stage IV Extrapulmonary Arm I (DD-4A, MVI); Stage IV Extrapulmonary Arm II (DD-4A, M); Stage IV Extrapulmonary Arm III (DD-4A, MVI); Stage IV Extrapulmonary Arm IV (DD-4A, M); Stage IV Extrapulmonary Arm IX (MVI); Stage IV Extrapulmonary Arm V (DD-4A, UH-3); Stage IV Extrapulmonary Arm VI (DD-4A, MVI); Stage IV Extrapulmonary Arm VII (DD-4A, M); Stage IV Extrapulmonary Arm VIII (UH-3); Stage IV Extrapulmonary Arm X (M); Stage IV Lung Metastases Arm I (DD-4A); Stage IV Lung Metastases Arm II (DD-4A, MVI); Stage IV Lung Metastases Arm III (DD-4A, MVI)
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
  Arms: Stage I, Arm IV (UH-3); Stage III, Arm II-Upfront/Delayed (DD-4A, UH-3); Stage III, Arm IIA (MVI); Stage III, Arm IIB (M); Stage III, Arm III-Upfront/Delayed (DD-4A, MVI); Stage III, Arm IV-Upfront/Delayed (DD-4A, M); Stage III, Arm IX-Upfront/Delayed (MVI); Stage III, Arm VB-Upfront/Delayed (M); Stage III, Arm VI-Upfront/Delayed (DD-4A, MVI); Stage III, Arm VII-Upfront/Delayed (DD-4A, M); Stage III, Arm VIII-Upfront/Delayed (UH-3); Stage III, Arm X-Upfront/Delayed (M); Stage IV Arm II-Upfront-Delayed (DD-4A, UH-3); Stage IV Arm III-Upfront-Delayed (DD-4A, MVI); Stage IV Arm IV-Upfront-Delayed (DD-4A, M); Stage IV Arm IX-Upfront-Delayed (MVI); Stage IV Arm VB-Upfront-Delayed (M); Stage IV Arm VI-Upfront-Delayed (DD-4A, MVI); Stage IV Arm VII-Upfront-Delayed (DD-4A, M); Stage IV Arm VIII-Upfront-Delayed (UH-3); Stage IV Arm X-Upfront-Delayed (M); Stage IV Extrapulmonary Arm I (DD-4A, MVI); Stage IV Extrapulmonary Arm II (DD-4A, M); Stage IV Extrapulmonary Arm III (DD-4A, MVI); Stage IV Extrapulmonary Arm IV (DD-4A, M); Stage IV Extrapulmonary Arm IX (MVI); Stage IV Extrapulmonary Arm V (DD-4A, UH-3); Stage IV Extrapulmonary Arm VI (DD-4A, MVI); Stage IV Extrapulmonary Arm VII (DD-4A, M); Stage IV Extrapulmonary Arm VIII (UH-3); Stage IV Extrapulmonary Arm X (M); Stage IV Lung Metastases Arm II (DD-4A, MVI); Stage IV Lung Metastases Arm III (DD-4A, MVI)
Drug: Irinotecan — Given IV
  Arms: Stage I, Arm IV (UH-3); Stage II, Arm II (EE-4A, VIVA); Stage III, Arm II-Upfront/Delayed (DD-4A, UH-3); Stage III, Arm IIA (MVI); Stage III, Arm III-Upfront/Delayed (DD-4A, MVI); Stage III, Arm IX-Upfront/Delayed (MVI); Stage III, Arm VI-Upfront/Delayed (DD-4A, MVI); Stage III, Arm VIII-Upfront/Delayed (UH-3); Stage IV Arm II-Upfront-Delayed (DD-4A, UH-3); Stage IV Arm III-Upfront-Delayed (DD-4A, MVI); Stage IV Arm IX-Upfront-Delayed (MVI); Stage IV Arm VI-Upfront-Delayed (DD-4A, MVI); Stage IV Arm VIII-Upfront-Delayed (UH-3); Stage IV Extrapulmonary Arm I (DD-4A, MVI); Stage IV Extrapulmonary Arm III (DD-4A, MVI); Stage IV Extrapulmonary Arm IX (MVI); Stage IV Extrapulmonary Arm V (DD-4A, UH-3); Stage IV Extrapulmonary Arm VI (DD-4A, MVI); Stage IV Extrapulmonary Arm VIII (UH-3); Stage IV Lung Metastases Arm II (DD-4A, MVI)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
  Arms: Stage I, Arm I (EE-4A); Stage I, Arm III (DD-4A); Stage I, Arm IV (UH-3); Stage II, Arm I (EE-4A); Stage II, Arm II (EE-4A, VIVA); Stage II, Arm III (EE-4A, DD-4A); Stage III, Arm I (DD-4A, EE-4A); Stage III, Arm I-Upfront/Delayed (DD-4A, EE-4A); Stage III, Arm II (DD-4A); Stage III, Arm II-Upfront/Delayed (DD-4A, UH-3); Stage III, Arm IIA (MVI); Stage III, Arm IIB (M); Stage III, Arm III-Upfront/Delayed (DD-4A, MVI); Stage III, Arm IV-Upfront/Delayed (DD-4A, M); Stage III, Arm IX-Upfront/Delayed (MVI); Stage III, Arm V-Upfront/Delayed (DD-4A); Stage III, Arm VA-Upfront/Delayed (DD-4A); Stage III, Arm VB-Upfront/Delayed (M); Stage III, Arm VI-Upfront/Delayed (DD-4A, MVI); Stage III, Arm VII-Upfront/Delayed (DD-4A, M); Stage III, Arm VIII-Upfront/Delayed (UH-3); Stage III, Arm X-Upfront/Delayed (M); Stage IV Arm I-Upfront-Delayed (DD-4A, EE-4A); Stage IV Arm II-Upfront-Delayed (DD-4A, UH-3); Stage IV Arm III-Upfront-Delayed (DD-4A, MVI); Stage IV Arm IV-Upfront-Delayed (DD-4A, M); Stage IV Arm IX-Upfront-Delayed (MVI); Stage IV Arm V-Upfront-Delayed (DD-4A); Stage IV Arm VA-Upfront-Delayed (DD-4A); Stage IV Arm VB-Upfront-Delayed (M); Stage IV Arm VI-Upfront-Delayed (DD-4A, MVI); Stage IV Arm VII-Upfront-Delayed (DD-4A, M); Stage IV Arm VIII-Upfront-Delayed (UH-3); Stage IV Arm X-Upfront-Delayed (M); Stage IV Extrapulmonary Arm I (DD-4A, MVI); Stage IV Extrapulmonary Arm II (DD-4A, M); Stage IV Extrapulmonary Arm III (DD-4A, MVI); Stage IV Extrapulmonary Arm IV (DD-4A, M); Stage IV Extrapulmonary Arm IX (MVI); Stage IV Extrapulmonary Arm V (DD-4A, UH-3); Stage IV Extrapulmonary Arm VI (DD-4A, MVI); Stage IV Extrapulmonary Arm VII (DD-4A, M); Stage IV Extrapulmonary Arm VIII (UH-3); Stage IV Extrapulmonary Arm X (M); Stage IV Lung Metastases Arm I (DD-4A); Stage IV Lung Metastases Arm II (DD-4A, MVI); Stage IV Lung Metastases Arm III (DD-4A, MVI)
Procedure: Nephrectomy — Undergo nephrectomy
  Arms: Stage III, Arm V-Upfront/Delayed (DD-4A); Stage IV Arm V-Upfront-Delayed (DD-4A)
Other: Patient Observation — Undergo observation after nephrectomy
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
  Arms: Stage I, Arm II (observation)
Procedure: Positron Emission Tomography — Undergo PET for patients with metastatic sites outside the chest/abdomen/pelvis documented during therapy
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
  Arms: Stage III, Arm IIA (MVI); Stage IV Arm VI-Upfront-Delayed (DD-4A, MVI); Stage IV Arm X-Upfront-Delayed (M); Stage IV Extrapulmonary Arm I (DD-4A, MVI); Stage IV Extrapulmonary Arm II (DD-4A, M); Stage IV Extrapulmonary Arm III (DD-4A, MVI); Stage IV Extrapulmonary Arm IV (DD-4A, M); Stage IV Extrapulmonary Arm IX (MVI); Stage IV Extrapulmonary Arm V (DD-4A, UH-3); Stage IV Extrapulmonary Arm VI (DD-4A, MVI); Stage IV Extrapulmonary Arm VII (DD-4A, M); Stage IV Extrapulmonary Arm VIII (UH-3); Stage IV Extrapulmonary Arm X (M)
Procedure: Ultrasound Imaging — Undergo ultrasound
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine
  Arms: Stage I, Arm I (EE-4A); Stage I, Arm III (DD-4A); Stage I, Arm IV (UH-3); Stage II, Arm I (EE-4A); Stage II, Arm II (EE-4A, VIVA); Stage II, Arm III (EE-4A, DD-4A); Stage III, Arm I (DD-4A, EE-4A); Stage III, Arm I-Upfront/Delayed (DD-4A, EE-4A); Stage III, Arm II (DD-4A); Stage III, Arm II-Upfront/Delayed (DD-4A, UH-3); Stage III, Arm IIA (MVI); Stage III, Arm IIB (M); Stage III, Arm III-Upfront/Delayed (DD-4A, MVI); Stage III, Arm IV-Upfront/Delayed (DD-4A, M); Stage III, Arm IX-Upfront/Delayed (MVI); Stage III, Arm V-Upfront/Delayed (DD-4A); Stage III, Arm VA-Upfront/Delayed (DD-4A); Stage III, Arm VI-Upfront/Delayed (DD-4A, MVI); Stage III, Arm VII-Upfront/Delayed (DD-4A, M); Stage III, Arm VIII-Upfront/Delayed (UH-3); Stage III, Arm X-Upfront/Delayed (M); Stage IV Arm I-Upfront-Delayed (DD-4A, EE-4A); Stage IV Arm II-Upfront-Delayed (DD-4A, UH-3); Stage IV Arm III-Upfront-Delayed (DD-4A, MVI); Stage IV Arm IV-Upfront-Delayed (DD-4A, M); Stage IV Arm IX-Upfront-Delayed (MVI); Stage IV Arm V-Upfront-Delayed (DD-4A); Stage IV Arm VA-Upfront-Delayed (DD-4A); Stage IV Arm VB-Upfront-Delayed (M); Stage IV Arm VI-Upfront-Delayed (DD-4A, MVI); Stage IV Arm VII-Upfront-Delayed (DD-4A, M); Stage IV Arm VIII-Upfront-Delayed (UH-3); Stage IV Arm X-Upfront-Delayed (M); Stage IV Extrapulmonary Arm I (DD-4A, MVI); Stage IV Extrapulmonary Arm II (DD-4A, M); Stage IV Extrapulmonary Arm III (DD-4A, MVI); Stage IV Extrapulmonary Arm IV (DD-4A, M); Stage IV Extrapulmonary Arm IX (MVI); Stage IV Extrapulmonary Arm V (DD-4A, UH-3); Stage IV Extrapulmonary Arm VI (DD-4A, MVI); Stage IV Extrapulmonary Arm VII (DD-4A, M); Stage IV Extrapulmonary Arm VIII (UH-3); Stage IV Extrapulmonary Arm X (M); Stage IV Lung Metastases Arm I (DD-4A); Stage IV Lung Metastases Arm II (DD-4A, MVI); Stage IV Lung Metastases Arm III (DD-4A, MVI)
Procedure: X-Ray Imaging — Undergo X-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase III trial studies using risk factors in determining treatment for children with favorable tissue (histology) Wilms tumors (FHWT). Wilms Tumor is the most common type of kidney cancer in children, and FHWT is the most common subtype. Previous large clinical trials have established treatment plans that are likely to cure most children with FHWT, however some children still have their cancer come back (called relapse) and not all survive. Previous research has identified features of FHWT that are associated with higher or lower risks of relapse. The term "risk" refers to the chance of the cancer coming back after treatment. Using results of tumor histology tests, biology tests, and response to therapy may be able to improve treatment for children with FHWT.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To maintain event-free survival (EFS) for Stage I favorable histology Wilms tumor (FHWT) patients without adverse biology who are also (1) 2 to < 4 years of age, OR (2) age < 2 years with tumor weight of 550 grams or more, OR (3) age 4+ years with epithelial histology subtype while reducing post-nephrectomy therapy from vincristine, actinomycin (EE-4A) to Nephrectomy Only. (Stage I Nephrectomy Only Stratum 2) II. To improve EFS for Stage I FHWT patients with age < 2 years AND nephrectomy weight < 550g AND whose tumors have adverse biology by treating with EE-4A instead of Nephrectomy Only. (Stage I EE-4A Stratum 3) III. To evaluate whether addition of vincristine and irinotecan to standard EE-4A (novel vincristine, actinomycin, irinotecan [Regimen VIVA]) is non-inferior to vincristine, actinomycin, doxorubicin (DD-4A) in terms of EFS among Stage II FHWT patients whose tumors demonstrate adverse biology. (Stage II: VIVA versus [vs] DD-4A Randomization) IV. To evaluate whether omission of doxorubicin (EE-4A) is non-inferior to historical DD-4A in Stage III FHWT patients with standard biology or post-therapy blastemal predominance. (Stage III: EE-4A) V. To demonstrate the non-inferiority of vincristine, actinomycin, doxorubicin, cyclophosphamide, etoposide and irinotecan (Regimen MVI) to vincristine, dactinomycin, doxorubicin, cyclophosphamide and etoposide (Regimen M) in the treatment of Stage III FHWT patients whose tumors exhibit adverse biology (post-chemotherapy blastemal predominance excluded). (Stage III: Regimen MVI vs Regimen M Randomization) VI. To demonstrate the non-inferiority of Regimen MVI to Regimen M in the treatment of Stage IV FHWT patients with adverse biology, slow incomplete lung response (SIR), or extrapulmonary metastases (EPM) (post-therapy blastemal predominance excluded). (Stage IV: Regimen MVI vs Regimen M Randomization) VII. To demonstrate the superiority of vincristine, doxorubicin, cyclophosphamide, etoposide, carboplatin and irinotecan (Regimen UH-3) vs historical DD-4A or Regimen M in treatment of Stage III or IV FHWT patients with blastemal predominance at delayed nephrectomy. (Stage III-IV: UH-3 [Blastemal Predominance])

SECONDARY OBJECTIVES:

I. To describe outcomes for Stage I FHWT patients without adverse biology who are either less than 4 years of age OR 4+ years of age with epithelial subtype who are treated with Nephrectomy Only and assess consistency with a matched historical control from the prior Children's Oncology Group (COG) therapeutic era. (Stage I: Nephrectomy Only) II. To describe outcomes for Stage I FHWT patients with adverse biology OR age > 4 and not epithelial subtype who are treated with post-nephrectomy EE-4A and assess consistency with a matched historical control from the prior COG therapeutic era. (Stage I: EE-4A) III. To describe overall survival in the cohort of modified very low risk (mVLR) patients who relapse following treatment with nephrectomy only and are assigned at relapse to DD-4A (if presumed or confirmed favorable histology Wilms tumor at relapse) or UH-3 (if evidence of anaplasia at relapse). (Stage I: Nephrectomy Only Relapse) IV. To describe outcomes for Stage II FHWT patients without adverse biology who are treated with post-nephrectomy EE-4A and assess consistency with a matched historical control from the prior COG therapeutic era. (Stage II: EE-4A) V. To compare outcomes of Stage II FHWT patients whose tumors are negative for combined loss of heterozygosity (LOH) but positive for 1q gain who are randomized to VIVA vs DD-4A on AREN2231 against historically matched patients treated with EE-4A during the prior COG therapeutic era. (Stage II VIVA vs DD-4A Stratum 1) VI. To compare outcomes of Stage II FHWT patients whose tumors are positive for combined LOH 1p AND 16q and who are randomized to VIVA vs DD-4A on AREN2231 against historically matched patients treated with DD-4A during the prior COG therapeutic era. (Stage II VIVA vs DD-4A Stratum 2) VII. To compare outcomes of Stage III FHWT patients whose tumors have adverse biology other than combined LOH and who are randomized to Regimen MVI vs Regimen M on AREN2231 against historically matched patients treated with DD-4A during the prior COG therapeutic era (post-chemotherapy blastemal predominance excluded). (Stage III Regimen MVI vs Regimen M Stratum 1) VIII. To compare outcomes of Stage III FHWT patients whose tumors have combined LOH and who are randomized to Regimen MVI vs Regimen M on AREN2231 against historically matched patients treated with Regimen M during the prior COG therapeutic era (post-chemotherapy blastemal predominance excluded). (Stage III Regimen MVI vs Regimen M Stratum 2) IX. To describe outcomes for Stage IV FHWT patients with rapid complete response of lung only metastases and no adverse biology who are treated with DD-4A on AREN2231 and assess consistency with a matched historical control from the prior COG therapeutic era (post-chemotherapy blastemal predominance excluded). (Stage IV: DD-4A) X. To compare outcomes of Stage IV lung only patients with either combined LOH 1p AND 16q or SIR who are randomized to Regimen MVI vs Regimen M on AREN2231 against historically matched patients treated with Regimen M during the prior COG therapeutic era (post-chemotherapy blastemal predominance excluded). (Stage IV Regimen MVI vs Regimen M Stratum 1) XI. To compare outcomes of Stage IV lung only rapid complete response (RCR) patients without combined LOH 1p AND 16q who are positive for other adverse biological factors and who are randomized to Regimen MVI vs Regimen M on AREN2231 against historically matched patients treated with DD-4A during the prior COG therapeutic era (post-chemotherapy blastemal predominance excluded). (Stage IV Regimen MVI vs Regimen M Stratum 2) XII. To compare outcomes of Stage IV patients with extrapulmonary metastases (EPM) who are randomized to Regimen MVI vs Regimen M on AREN2231 against historically matched patients treated with Regimen M during the prior COG therapeutic era (post-chemotherapy blastemal predominance excluded). (Stage IV Regimen MVI vs Regimen M Stratum 3) XIII. To report a pooled comparison of Regimen MVI vs Regimen M in Stage III or Stage IV randomized patients. (Stage III-IV Regimen MVI vs Regimen M) XIV. To compare outcomes of Stage III or IV FHWT patients with blastemal predominance at delayed nephrectomy who are treated with Regimen UH-3 on AREN2231 vs a historically matched cohort that received DD-4A in the prior COG therapeutic era. (Stage III-IV UH-3 Stratum 1) XV. To compare outcomes of Stage III or IV FHWT patients with blastemal predominance at delayed nephrectomy who are treated with Regimen UH-3 on AREN2231 vs a historically matched cohort that received Regimen M in the prior COG therapeutic era. (Stage III-IV UH-3 Stratum 2) XVI. To describe outcomes of Stage III or IV FHWT patients with delayed nephrectomy occurring after the start of Cycles 3 or 4 (super delayed) who are assigned to Regimen M or continued DD4A. (Stage III-IV Super Delayed Nephrectomy)

EXPLORATORY OBJECTIVES:

I. To determine the impact of imaging schedule and modality (chest x-ray [CXR], ultrasound [US], versus computed tomography/magnetic resonance imaging [CT/MRI], versus clinical symptoms) on relapse, timing of detection of relapse, burden of disease at relapse (as assessed by retrospective central imaging review), as well as impact on survival.

II. To analyze the impact of radiologically determined pulmonary tumor burden on outcomes.

III. To assess whether imaging modality (ultrasound, CT, MRI with or without hepatocyte specific contrast agent) at diagnosis is associated with detection of increased number of liver metastases, and whether modality choice impacts surgery and/or radiation planning for liver metastases.

IV. To accurately describe the responses of extrapulmonary metastases to the various therapeutic modalities (chemotherapy, radiation therapy, and surgery) through central review of institutional imaging at various stages of treatment, and to correlate institutionally interpreted radiologic response interpretations with central review.

V. To describe the association of the number of anatomically relevant and pathologically confirmed lymph nodes sampled and percent of positive lymph nodes (LNs) on EFS and overall survival (OS).

VI. To document the surgical and/or medical rationale and approach for biopsy (including type of biopsy, number of biopsies, and site of biopsy) for all patients who are treated with the approach of initial biopsy and delayed nephrectomy.

VII. To describe sites of recurrence for patients with liver metastases according to the surgery and/or radiation therapy administered for residual liver lesions at Week 6 and 12.

VIII. To increase the number of patients eligible to avoid lung radiation therapy (RT) by encouraging resection of residual pulmonary nodules for patients defined as Stage IV FHWT with standard biology and who have 1-3 residual pulmonary nodules on imaging after Cycle 2, by omitting lung RT for those who are found to have no viable tumor in resected nodules.

IX. To describe whether residual lung lesions at end of therapy are associated with relapse.

X. To improve the reliability of data derived from central surgical review through the implementation of a standardized operative note.

XI. To describe the treatment, perioperative morbidity and outcome of patients noted to have inferior vena cava (IVC) tumor thrombus at time of diagnosis, including surgical approach, pathology findings and specific radiation therapy received.

XII. To determine the feasibility of employing intensity modulated radiation therapy (IMRT) and proton therapy with central quality assurance (QA) monitoring within the prescribed time frame.

XIII. To determine the lung tumor and liver tumor control rate using IMRT and/or proton therapy and compare it to standard 3-dimensional radiotherapy in the current study and the AREN0533 study.

XIV. To determine the flank and abdominal tumor control rates in children with Stage IV FHWT who received abdominal radiotherapy after 2 cycles of chemotherapy in this study (delayed abdominal radiation) and compare it to AREN0533 study where abdominal radiotherapy was performed within 2 weeks of nephrectomy (upfront abdominal radiation).

XV. To compare abdominal relapse according to protocol-recommended radiotherapy fields (flank vs. whole abdominal) in the current study and compare it to the abdominal relapse according to radiotherapy fields (flank vs. whole abdominal) in the AREN0532 and AREN0533 studies.

XVI. To determine the impact of radiotherapy on local and distant control rates for EPM sites and compare them to EPM sites not receiving radiation.

XVII. To describe the rate and severity of recurrent hepatotoxicity in patients who undergo re-introduction of chemotherapy after experiencing hepatopathy.

XVIII. To collect serial blood and urine samples to bank for future research studies.

OUTLINE:

STAGE I FHWT: Patients will have already undergone nephrectomy and lymph node sampling prior to trial enrollment. Patients < 4 years old at diagnosis or with epithelial subtype FHWT of any age, undergo observation until tumor biomarker testing returns. Patients with adverse biology are assigned to Arm I. Patients with standard biology are assigned to Arm II and undergo observation post-nephrectomy until disease relapse. At the time of disease relapse, patients with favorable histology are assigned to Arm III, and patients with unfavorable (anaplastic) histology are assigned to Arm IV. Patients ≥ 4 years of age at diagnosis without epithelial FHWT are assigned to Arm I regardless of biology results.

* ARM I: Patients receive regimen EE-4A: Dactinomycin intravenously (IV) over 1-5 or 10-15 minutes on day 1 of cycles 1-7 and vincristine IV on days 1, 8, & 15 of cycles 1-3 and day 1 of cycles 4-7. Treatment repeats every 21 days for 7 cycles in the absence of disease progression or unacceptable toxicity.
* ARM II: Patients undergo observation without chemotherapy on study with ultrasounds and x-rays.
* ARM III: Patients receive regimen DD-4A: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycles 1, 3, 5, 7, & 9, vincristine IV on days 1, 8, & 15 of cycles 1-3 and day 1 of cycles 4-9, doxorubicin IV over 3-15 minutes on day 1 of cycles 2, 4, 6, & 8. Treatment repeats every 21 days for 9 cycles in the absence of disease progression or unacceptable toxicity.
* ARM IV: Patients receive regimen UH-3: Vincristine IV on days 1, 8, & 15 of cycles 1, 5, 7, 10, & 13, and days 1 & 8 of cycles 3, 4, 8, & 11, doxorubicin IV 3-15 minutes on day 1 of cycles 1, 5, 7, 10, & 13, cyclophosphamide IV over 30-60 minutes on day 1 of cycles 1, 5, 7, 10, & 13, and days 1-4 of cycles 2, 6, 9, 12, & 14, carboplatin IV over 15-60 minutes on day 1 of cycles 2, 6, 9, 12, and 14, etoposide IV over 60-120 minutes on days 1-4 of cycles 2, 6, 9, 12, & 14, and irinotecan IV over 90 minutes on days 1-5 of cycles 3, 4, 8, & 11. Treatment repeats every 21 days for 14 cycles in the absence of disease progression or unacceptable toxicity.

STAGE II FHWT: Patients receive one cycle of regimen EE-4A as in STAGE I FHWT Arm I. Patients with standard biology are assigned to Arm I below. Patients with adverse biology are randomized to Arm II or Arm III below.

* ARM I: Patients receive cycles 2-7 of regimen EE-4A as in STAGE I FHWT Arm I.
* ARM II: Patients receive cycles 2-9 of regimen VIVA: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycles 3, 5, 7, & 9, vincristine IV on days 1, 8, & 15 of cycles 2-3 and day 1 of cycles 4-9, irinotecan IV over 90 minutes daily on days 1-5 of cycles 2, 4, 6, & 8. Treatment repeats every 21 days for 8 cycles in the absence of disease progression or unacceptable toxicity.
* ARM III: Patients receive cycles 2-9 of regimen DD-4A: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycles 3, 5, 7, and 9, vincristine IV on days 1, 8, and 15 of cycles 2-3 and day 1 of cycles 4-9, and doxorubicin IV over 3-15 minutes on day 1 of cycles 2, 4, 6, & 8. Treatment repeats every 21 days for 8 cycles in the absence of disease progression or unacceptable toxicity.

STAGE III FHWT: Patients able to undergo an upfront nephrectomy receive cycle 1 treatment of regimen DD-4A: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycles 1, 3, 5, 7, & 9, vincristine IV on days 1, 8, & 15 of cycles 1-3 and day 1 of cycles 4-9, doxorubicin IV over 3-15 minutes on day 1 of cycles 2, 4, 6, & 8. Patients with standard biology are assigned to Arm I below. Patients with adverse biology are assigned to Arm II below.

* ARM I: Patients receive cycles 2-7 of regimen EE-4A as in STAGE I FHWT Arm I.
* ARM II: Patients receive cycle 2 treatment of regimen DD-4A as in STAGE II FHWT Arm III above. They are then randomized to Arm IIA or Arm IIB below.

  * ARM IIA: Patients receive regimen MVI: Vincristine IV on days 1, 8, & 15 of cycle 3, days 8 & 15 of cycle 4, and day 1 of cycles 5 & 7-13, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycles 3, 7, 9, 11, & 13, doxorubicin IV over 3-15 minutes on day 1 of cycles 3, 7, 9, 11, & 13, cyclophosphamide IV over 15-30 minutes daily on days 1-5 of cycles 4 and 6, irinotecan IV over 90 minutes daily on days 1-5 of cycles 5, 8, 10 & 12, and etoposide IV over 60-120 minutes daily on days 1-5 of cycles 4 and 6. Treatment repeats every 21 days for 11 cycles in the absence of disease progression or unacceptable toxicity.
  * ARM IIB: Patients receive regimen M: Cyclophosphamide IV over 15-30 minutes daily on days 1-5 of cycles 3, 4, 7, & 9, etoposide IV over 60-120 minutes daily on days 1-5 of cycles 3, 4, 7, & 9, vincristine IV on days 8 & 15 of cycles 3 & 4 and day 1 of cycles 5, 6, 8, 10, & 11, dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycles 5, 6, 8, 10, & 11, and doxorubicin IV over 3-15 minutes of cycles 5, 6, 8, 10, & 11. Treatment repeats every 21 days for 9 cycles in the absence of disease progression or unacceptable toxicity.

STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY): Patients receive cycles 1-2 of regimen DD-4A: Dactinomycin IV over 1-5 or 10-15 minutes on day 1 of cycle 1, vincristine IV on days 1, 8, and 15 of cycles 1-2, and doxorubicin IV over 3-15 minutes on day 1 of cycle 2. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity.

* PATIENTS ABLE TO UNDERGO A DELAYED NEPHRECTOMY AFTER CYCLE 2: Patients with standard biology and low or intermediate risk histology are assigned to Arm I below. Patients with high risk histology are assigned to Arm II below. Patients with adverse biology and low or intermediate risk histology are randomized to Arm III or Arm IV below.
* PATIENTS UNABLE TO UNDERGO A DELAYED NEPHRECTOMY AFTER CYCLE 2: Patients with standard biology are assigned to Arm V below. Patients with adverse biology are randomized to Arm VI or Arm VII below.
* ARM I: Patients receive cycles 3-7 of regimen EE-4A as in STAGE I FHWT Arm I above.
* ARM II: Patients receive regimen UH-3 as in STAGE I FHWT Arm IV above: Vincristine IV on days 1, 8, & 15 of cycles 1, 5, 7, 10, & 13, and days 1 & 8 of cycles 3, 4, 8, & 11, doxorubicin IV 3-15 minutes on day 1 of cycles 1, 5, 7, 10, & 13, cyclophosphamide IV over 30-60 minutes on day 1 of cycles 1, 5, 7, 10, & 13, and days 1-4 of cycles 2, 6, 9, 12, & 14, carboplatin IV over 15-60 minutes on day 1 of cycles 2, 6, 9, 12, and 14, etoposide IV over 60-120 minutes on days 1-4 of cycles 2, 6, 9, 12, & 14, and irinotecan IV over 90 minutes on days 1-5 of cycles 3, 4, 8, & 11. Treatment repeats every 21 days for 14 cycles in the absence of disease progression or unacceptable toxicity.
* ARM III: Patients receive regimen MVI as in STAGE III FHWT Arm IIA above.
* ARM IV: Patients receive regimen M as in STAGE III FHWT Arm IIB above.
* ARM V: Patients receive cycles 3-4 of regimen DD-4A as in STAGE II FHWT Arm III above. They then undergo delayed nephrectomy after cycle 3 or 4. Patients with low or intermediate risk histology who still have standard biology are then assigned to Arm VA. Patients with low or intermediate risk histology with new adverse biology (positive lymph nodes, and LOH of 1p or 16q from original biopsy) are then assigned to Arm VB. Patients with high risk histology are assigned to Arm VIII below.

  * ARM VA: Patients receive cycles 5-9 (or 4-9 if nephrectomy occurred after cycle 3) of regimen DD-4A as in STAGE II FHWT Arm III above.
  * ARM VB: Patients receive cycles 5-9 (or 4-9 if nephrectomy occurred after cycle 3) of regimen M as in STAGE III FHWT Arm IIB above.
* ARM VI: Patients receive cycles 3-4 of regimen MVI as in STAGE III FHWT Arm IIA above. Patients with high risk histology after delayed nephrectomy after cycle 3 or 4 are assigned to Arm VIII. Patients with low or intermediate risk histology after delayed nephrectomy after cycle 3 or 4 are assigned to Arm IX.
* ARM VII: Patients receive cycles 3-4 of regimen M as in STAGE III FHWT Arm IIB above. Patients with high risk histology after delayed nephrectomy after cycle 3 or 4 are assigned to Arm VIII. Patients with low or intermediate risk histology after delayed nephrectomy after cycle 3 or 4 are assigned to Arm X.
* ARM VIII: Patients receive regimen UH-3 as in STAGE I FHWT Arm IV above.
* ARM IX: Patients receive cycles 5-13 (or 4-13 if nephrectomy occurred after cycle 3) of regimen MVI as in STAGE III FHWT Arm IIA above.
* ARM X: Patients receive cycles 5-11 (or 4-11 if nephrectomy occurred after cycle 3) of regimen M as in STAGE III FHWT Arm IIB above.

STAGE IV FHWT LUNG METASTASES (UPFRONT NEPHRECTOMY): Patients receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above. Patients with standard biology and rapid complete lung response (RCR) are assigned to Arm I below. Patients with standard biology and slow incomplete lung response (SIR), or adverse biology (with either RCR or SIR) are randomized to Arm II or Arm III below.

* ARM I: Patients receive cycles 3-9 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) Arms V and VA above.
* ARM II: Patients receive regimen MVI as in STAGE III FHWT Arm IIA above.
* ARM III: Patients receive regimen M as in STAGE III FHWT Arm IIB above.

STAGE IV FHWT LUNG METASTASES (UPFRONT BIOPSY/DELAYED NEPHRECTOMY): Patients receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above.

* PATIENTS ABLE TO UNDERGO A DELAYED NEPHRECTOMY AFTER CYCLE 2: Patients with standard biology, low or intermediate risk histology, and RCR are assigned to Arm I below. Patients with high risk histology are assigned to Arm II below. Patients with adverse biology OR SIR and low or intermediate risk histology are randomized to Arm III or Arm IV below.
* PATIENTS UNABLE TO UNDERGO A DELAYED NEPHRECTOMY AFTER CYCLE 2: Patients with standard biology and RCR are assigned to Arm V below. Patients with standard biology and SIR OR adverse biology and either SIR or RCR are randomized to Arm VI or Arm VII below.
* ARM I: Patients receive cycles 3-7 of regimen EE-4A as in STAGE I FHWT Arm I above.
* ARM II: Patients receive regimen UH-3 as in STAGE I FHWT Arm IV above.
* ARM III: Patients receive regimen MVI as in STAGE III FHWT Arm IIA above.
* ARM IV: Patients receive regimen M as in STAGE III FHWT Arm IIB above.
* ARM V: Patients receive cycles 3-4 of regimen DD-4A as in STAGE II FHWT Arm II above. They then undergo delayed nephrectomy after cycle 3 or 4. Patients with low or intermediate risk histology still with standard biology are then assigned to Arm VA. Patients with low or intermediate risk histology and new adverse biology (positive lymph nodes, and LOH of 1p or 16q from original biopsy) are then assigned to Arm VB. Patients with high risk histology are assigned to Arm VIII below.

  * ARM VA: Patients receive cycles 5-9 (or 4-9 if nephrectomy occurred after cycle 3) of regimen DD-4A as in STAGE II FHWT Arm II above.
  * ARM VB: Patients receive regimen M as in STAGE III FHWT Arm IIB above.
* ARM VI: Patients receive cycles 3-4 of regimen MVI as in STAGE III FHWT Arm IIA above. Patients with high risk histology after delayed nephrectomy in cycle 3 or 4 are assigned to Arm VIII. Patients with low or intermediate risk histology after delayed nephrectomy in cycle 3 or 4 are assigned to Arm IX.
* ARM VII: Patients receive cycles 3-4 of regimen M as in STAGE III FHWT Arm IIB above. Patients with high risk histology after delayed nephrectomy in cycle 3 or 4 are assigned to Arm VIII. Patients with low or intermediate risk histology after delayed nephrectomy in cycle 3 or 4 are assigned to Arm X.
* ARM VIII: Patients receive regimen UH-3 as in STAGE I FHWT Arm IV above.
* ARM IX: Patients receive cycles 5-13 (or 4-13 if nephrectomy occurred after cycle 3) of regimen MVI as in STAGE III FHWT Arm IIA above.
* ARM X: Patients receive cycles 5-11 (or 4-11 if nephrectomy occurred after cycle 3) of regimen M as in STAGE III FHWT Arm IIB above. NOTE: Patients who receive 4 cycles of initial treatment per regimen DD-4A omit cycle 11.

STAGE IV FHWT EXTRAPULMONARY METASTASES: Patients receive cycles 1-2 of regimen DD-4A as in STAGE III FHWT (UPFRONT BIOPSY/DELAYED NEPHRECTOMY) above.

PATIENTS ABLE TO UNDERGO UPFRONT NEPHRECTOMY: Patients are randomized to Arm I or II below.

PATIENTS ABLE TO UNDERGO DELAYED NEPHRECTOMY AFTER CYCLE 2: Patients with low or intermediate risk histology are randomized to Arm III or IV.

PATIENTS ABLE TO UNDERGO DELAYED NEPHRECTOMY AFTER CYCLE 2: Patients with high risk histology are assigned to Arm V.

PATIENTS UNABLE TO UNDERGO DELAYED NEPHRECTOMY AFTER CYCLE 2: Patients are randomized to Arm VI or VII.

* ARM I: Patients receive regimen MVI as in STAGE III FHWT Arm IIA above.
* ARM II: Patients receive regimen M as in STAGE III FHWT Arm IIB above.
* ARM III: Patients receive regimen MVI as in STAGE III FHWT Arm IIA above.
* ARM IV: Patients receive regimen M as in STAGE III FHWT Arm IIB above.
* ARM V: Patients receive regimen UH-3 as in STAGE I FHWT Arm IV above.
* ARM VI: Patients receive cycles 3-4 of regimen MVI as in STAGE III FHWT Arm IIA above. Patients undergoing nephrectomy after cycles 3 or 4 and with low or intermediate risk histology are assigned to Arm IX below. Patients undergoing nephrectomy after cycles 3 or 4 and with high risk histology are assigned to Arm VIII below
* ARM VII: Patients receive cycles 3-4 of regimen M as in STAGE III FHWT Arm IIB above. Patients undergoing nephrectomy after cycles 3 or 4 and with low or intermediate risk histology are assigned to Arm X below. Patients undergoing nephrectomy after cycles 3 or 4 and with high risk histology are assigned to Arm VIII below.
* ARM VIII: Patients receive regimen UH-3 as in STAGE I FHWT Arm IV above.
* ARM IX: Patients receive cycles 5-13 (or 4-13 if nephrectomy occurred after cycle 3) of regimen MVI as in STAGE III FHWT Arm IIA above.
* ARM X: Patients receive cycles 5-11 (or 4-11 if nephrectomy occurred after cycle 3) of regimen M as in STAGE III FHWT Arm IIB above.

  * NOTE: Patients receiving regimens EE-4A, DD-4A, VIVA, M, MVI & UH3 also undergo computed tomography (CT), CT or magnetic resonance imaging (MRI), ultrasound, and X-ray imaging throughout the trial. Patients with metastatic sites outside the chest/abdomen/pelvis documented during therapy may also undergo bone scan and/or positron emission tomography (PET).

After completion of study treatment, patients are followed for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be enrolled on APEC14B1 and consent to Part A - Eligibility Screening prior to enrollment on AREN2231.
* Patients must be < 30 years old at enrollment.
* Patients with newly diagnosed Stage I-IV Favorable Histology Wilms Tumor confirmed by central review and with a qualifying Initial Stratum Assignment on APEC14B1.
* Patients must receive a qualifying Initial Stratum Assignment on APEC14B1-REN by Day 14 post-diagnostic procedure (nephrectomy or biopsy), where that procedure is Day 0.

  * Patients must enroll on AREN2231 by Day 14.
  * Exceptions: If patient reaches Day 14 (post initial diagnostic nephrectomy or biopsy) without receiving an Initial Stratum Assignment on APEC14B1-REN, patient will not be eligible for enrollment on AREN2231 unless all required materials (reports and Case Report Forms and specimens) for an Initial Stratum Assignment arrived by Day 7, but an Initial Stratum Assignment was not completed by Day 14. In these circumstances, after obtaining appropriate protocol consent, the patient may proceed with treatment according to local institutional staging and enroll within 5 calendar days of notification of the central Initial Stratum Assignment being issued, only if the AREN2231 Initial Stratum Assignment is in agreement with any treatment already initiated. If the Initial Stratum Assignment is not in agreement with the local institution's assessment then the patient will be ineligible for AREN2231.
* All sites must have sent or plan to send diagnostic tumor sample for molecular testing through a Clinical Laboratory Improvement Act (CLIA)-certified (or equivalent if outside of the United States [US]) laboratory that can detect Loss of Heterozygosity (LOH) of chromosome 1p AND 16q, and gain of chromosome 1q. Patients potentially eligible for mVLR must also have LOH of chromosome 11p15 included.

  * Note: Patients are eligible for enrollment prior to obtaining these molecular testing results, and it is strongly recommended that patients are enrolled before these results are available. However, molecular results must be returned and uploaded to APEC14B1-REN for integration into risk stratification by the required timepoints (specific timelines vary by treatment arm). Patients who do not have molecular results available by the arm-specific timepoints may be taken off protocol therapy.
* Patients who have an upfront nephrectomy must have at least one lymph node sampled and confirmed as a lymph node by central pathology review to be eligible.

  * Note: Lymph node sampling will also be required at delayed nephrectomy. Patients who do not have a lymph node sampled and confirmed as a lymph node by central pathology review at delayed nephrectomy will be taken off protocol therapy.
* Karnofsky performance status must be ≥ 50 for patients > 16 years of age and the Lansky performance status must be ≥ 50 for patients ≤ 16 years of age.
* Serum total bilirubin ≤ 1.5 X upper limit of normal (ULN) OR direct bilirubin ≤ 3X ULN for subjects with total bilirubin levels > 1.5 ULN (within 7 days prior to enrollment).
* Aspartate aminotransferase (AST/serum glutamate oxaloacetic transaminase [SGOT]) OR alanine transaminase (ALT/serum glutamic pyruvate transaminase [SGPT]) ≤ 3X ULN OR ≤ 5 X ULN for patients with liver metastases (within 7 days prior to enrollment).
* Shortening fraction of ≥ 27% by echocardiogram, or ejection fraction of ≥ 50% (within 7 days prior to enrollment)

  * Note: This criteria only applies to patients centrally classified as Stage IV. Stage II and III patients subsequently assigned to a doxorubicin arm will be off protocol therapy if they do not meet this criteria at time of cardiac function assessment.
* Known HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* All patients and/or their parents or legal guardians must sign a written informed consent.
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met.

Exclusion Criteria:

* Patient with a diagnosis of Stage V Bilateral Wilms Tumor.
* Patients who in the opinion of the investigator are not able to comply with the study procedures are not eligible.
* Patients with any uncontrolled, intercurrent illness including but not limited to symptomatic congestive heart failure.
* Patients with Stage I FHWT with a known or suspected Wilms Tumor predisposition syndrome or condition (contralateral nephrogenic rests and/or unilateral multicentric tumors) are excluded from treatment on the mVLR (Nephrectomy Only) arm.

  * Notes:

    * In the context of the renal tumor protocols, multicentric tumors and multifocal tumors are equivalent terms, and refer to the occurrence of two or more tumors arising within one kidney.
    * Exclusion from the Nephrectomy Only arm applies to two groups of patients:

      * Patients < 4 years with Stage I FHWT other than epithelial subtype AND
      * Stage I patients of any age with Epithelial WT
    * For the purpose of exclusion from the Nephrectomy Only Arm, known or suspected WT predisposition syndromes or conditions are defined as follows:

      * WT Predisposition Syndromes: Beckwith Wiedemann Spectrum, Denys Drash, Trisomy 18, Idiopathic Hemihypertrophy/Isolated Lateralized Overgrowth, WAGR, Simpson-Golabi-Behmel, Bohring-Opitz, or other conditions considered by treating physician to predispose to WT.
      * WT Predisposing Conditions:

        * A unilateral WT and (radiologic or pathologic) determination of contralateral nephrogenic rest(s) AND/OR
        * Unilateral multicentric WT
* Patients treated with partial nephrectomy at initial diagnosis are excluded from mVLR (Nephrectomy Only) arm.
* Patients with lung metastases as the only metastatic site who already had complete resection of all radiologically evident lung nodules, and have at least one nodule confirmed pathologically as tumor.

  * Please note: Those with lung metastases as the only metastatic site who have complete resection of all radiologically evident lung nodules after enrollment but prior to the lung imaging following Cycle 2 of DD-4A will be inevaluable for lung assessment and subsequent stratum assignment and will, therefore, come off protocol therapy.
* Patients with known Charcot-Marie-Tooth syndrome.
* Patients who have had prior tumor-directed chemotherapy or radiotherapy for the current diagnosis except for therapy delivered for an emergent issue, as medically indicated.
* Patients who will potentially require doxorubicin on this study and have previously received doxorubicin for another diagnosis.
* Patients receiving concurrent chemotherapy for a different diagnosis.
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential.
* Lactating females who plan to breastfeed their infants.
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1656 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2031-02-13 (Estimated); Study Completion 2031-02-13 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Up to 4 years from study entry
  Kaplan-Meier method will be used to estimate 4-year EFS, defined as the time from randomization or first diagnostic nephrectomy or biopsy until relapse or disease progression, secondary malignancy, or death.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 4 years from study entry
  Kaplan-Meier method will be used to estimate 4-year OS, defined as the time from randomization or first diagnostic nephrectomy or biopsy until relapse or disease progression, secondary malignancy, or death

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Mullen, Principal Investigator — Children's Oncology Group
Locations (148):
- United States (136):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (12):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec